CLINICAL TRIAL: NCT06241235
Title: A Phase I/II Study to Evaluate Safety and Pharmacokinetics and Initial Efficacy of ZG005 in Combination With Paclitaxel Plus Cisplatin/Carboplatin ± Bevacizumab in Patients With Advanced Cervical Carcinoma
Brief Title: Study of ZG005 in Combination With Paclitaxel＋Platinum-based ± Bevacizumab in Patients With Advanced Cervical Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZG005-003
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Injections; Paclitaxel; Bevacizumab; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Part 1 is a dose escalation study of ZG005 combined with paclitaxel and platinum-based ± bevacizumab to evaluate the tolerability and safety of the combination regimen
  Interventions: Drug: ZG005 Powder for Injection; Drug: Paclitaxel; Biological: Bevacizumab; Drug: Cisplatin; Drug: Carboplatin
- Part 2: Dose Expansion (Experimental): Part 2 is a dose expansion study to further evaluate the initial efficacy and safety of the combination regimen
  Interventions: Drug: ZG005 Powder for Injection; Drug: Paclitaxel; Biological: Bevacizumab; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: ZG005 Powder for Injection — ZG005 for dose escalations are set as 10 mg/kg, 15 mg/kg and other doses after discussion, intravenous infusion(IV), once every 3 weeks (Q3W). ZG005 for dose-expansion stage will commence after the Recommended Phase 2 Dose (RP2D) is determined during the dose-escalation stage.
  Other Names: ZG005
Drug: Paclitaxel — IV infusion
Biological: Bevacizumab — IV infusion
Drug: Cisplatin — IV infusion
Drug: Carboplatin — IV infusion

SUMMARY:
This is a multicenter, open-label phase I/II study for the first-line treatment of advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form.
* Female 18-70 years of age;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or
* Life expectancy ≥ 3 months.

Exclusion Criteria:

* Patients were deemed unsuitable for participating in the study by the investigator for any reasons.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Up to 2 years
Objective Response Rate (ORR) | Up to 2 years
  ORR was defined as the percentage of the participants in the analysis population who have a Complete Response or a Partial Response. The ORR per RECIST 1.1 as assessed by Investigator is presented.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Zhejiang Cancer Hospital, Zhejiang, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No